CLINICAL TRIAL: NCT02799641
Title: Double-blind, Randomized, Placebo-controlled Study on the Effect of Multimodal Analgesia on Pain With Insertion of Levonorgestrel-releasing Intrauterine System
Brief Title: Effect of Multimodal Analgesia on Pain With Insertion of Levonorgestrel-releasing IUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-062
Record Dates: First submitted 2015-10-28; First posted 2016-06-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Contraception
Keywords: Contraception; IUD; levonorgestrel releasing intrauterine device; lidocaine; valium; diazepam; pain; VAS; visual analog scale
MeSH Terms: conditions — Pain | interventions — Diazepam; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Control arm receives ibuprofen, placebo pill, and placebo injection.
  Interventions: Other: Placebo pill; Other: Placebo injection
- Treatment (Experimental): Treatment arm receives ibuprofen, diazepam pill, and lidocaine injection.
  Interventions: Drug: Diazepam; Drug: Lidocaine

INTERVENTIONS:
Drug: Diazepam — 5 mg Diazepam
  Other Names: Valium
  Arms: Treatment
Drug: Lidocaine — 2 ml of 2% lidocaine
  Other Names: Xylocaine
  Arms: Treatment
Other: Placebo pill — Placebo pill
  Arms: Control
Other: Placebo injection — Placebo injection
  Arms: Control

SUMMARY:
Does the addition of cervical lidocaine injections and valium to the current practice result in decreased reported pain with tenaculum placement, IUD insertion, and post procedural discomfort? The current practice is ibuprofen alone or no medication.

DETAILED DESCRIPTION:
Long acting reversible contraception, including intrauterine devices (IUDs), provide birth control for an extended period of time. IUDs are the most effective type of reversible birth control for women who do not wish to become pregnant over the next couple years, have the lowest failure rate (Winner, 2012), and in 2007, were used by more than 180 million women worldwide (Darney, 2010). Despite the high efficacy and low rates of side effects, women may decline placement of an IUD due to fear of pain associated with placement. IUDs may act as a barrier to women selecting this method of contraception. Currently there is no consensus in the literature as to the most effective way to address analgesia surrounding IUD insertion.

In order to eliminate barriers to selecting the IUD for contraception, improve the experience of women undergoing placement, and standardize local practices, investigators want to investigate analgesic options affecting patients' perception of pain during the various steps of IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Desires to undergo placement of a levonorgestrel containing intrauterine device

Exclusion Criteria:

* Device manufacturer contraindications such as signs of genital infection, positive urine pregnancy test, abnormal vaginal bleeding, abnormal sized uterus that sounds <6cm or >10cm, and all other contraindications to placement of a levonorgestrel containing IUD.
* Patients with a history of drug abuse.
* History of a prior IUD
* Current use of medications for anxiety
* Also, a diagnosis of chronic pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-07; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analog Score) pain score | At IUD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth Inc.
Locations (1):
- Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero L, Pazol K, Warner L, Gavin L, Moskosky S, Besera G, Loyola Briceno AC, Jatlaoui T, Barfield W; Centers for Disease Control and Prevention (CDC). Vital signs: trends in use of long-acting reversible contraception among teens aged 15-19 years seeking contraceptive services-United States, 2005-2013. MMWR Morb Mortal Wkly Rep. 2015 Apr 10;64(13):363-9. PMID 25856258
- [Background] Li R, Ruckle HC, Creech JD, Culpepper DJ, Lightfoot MA, Alsyouf M, Nicolay L, Jellison F, Baldwin DD. A prospective, randomized, controlled trial assessing diazepam to reduce perception and recall of pain during transrectal ultrasonography-guided biopsy of the prostate. J Endourol. 2014 Jul;28(7):881-6. doi: 10.1089/end.2014.0043. Epub 2014 May 5. PMID 24641687
- [Background] Pergialiotis V, Vlachos DG, Protopappas A, Vlachos GD. Analgesic options for placement of an intrauterine contraceptive: a meta-analysis. Eur J Contracept Reprod Health Care. 2014 Jun;19(3):149-60. doi: 10.3109/13625187.2014.903238. Epub 2014 May 14. PMID 24828514
- [Background] Ekelund M, Melander M, Gemzell-Danielsson K. Intrauterine contraception: attitudes, practice, and knowledge among Swedish health care providers. Contraception. 2014 May;89(5):407-12. doi: 10.1016/j.contraception.2013.12.014. Epub 2014 Jan 7. PMID 24485096
- [Background] Goldthwaite LM, Baldwin MK, Page J, Micks EA, Nichols MD, Edelman AB, Bednarek PH. Comparison of interventions for pain control with tenaculum placement: a randomized clinical trial. Contraception. 2014 Mar;89(3):229-33. doi: 10.1016/j.contraception.2013.11.018. Epub 2013 Dec 10. PMID 24405796
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Scavuzzi A, Souza AS, Costa AA, Amorim MM. Misoprostol prior to inserting an intrauterine device in nulligravidas: a randomized clinical trial. Hum Reprod. 2013 Aug;28(8):2118-25. doi: 10.1093/humrep/det240. Epub 2013 Jun 5. PMID 23739219
- [Background] Ibrahim ZM, Sayed Ahmed WA. Sublingual misoprostol prior to insertion of a T380A intrauterine device in women with no previous vaginal delivery. Eur J Contracept Reprod Health Care. 2013 Aug;18(4):300-8. doi: 10.3109/13625187.2013.800855. Epub 2013 Jun 10. PMID 23751152
- [Background] Waddington A, Reid R. More harm than good: the lack of evidence for administering misoprostol prior to IUD insertion. J Obstet Gynaecol Can. 2012 Dec;34(12):1177-1179. doi: 10.1016/S1701-2163(16)35465-2. PMID 23231800
- [Background] Rossi V, Pourtois G. Transient state-dependent fluctuations in anxiety measured using STAI, POMS, PANAS or VAS: a comparative review. Anxiety Stress Coping. 2012 Nov;25(6):603-45. doi: 10.1080/10615806.2011.582948. Epub 2011 Aug 10. PMID 21827372
- [Background] Polyzos NP, Zavos A, Valachis A, Dragamestianos C, Blockeel C, Stoop D, Papanikolaou EG, Tournaye H, Devroey P, Messinis IE. Misoprostol prior to hysteroscopy in premenopausal and post-menopausal women. A systematic review and meta-analysis. Hum Reprod Update. 2012 Jul;18(4):393-404. doi: 10.1093/humupd/dms014. Epub 2012 Apr 27. PMID 22544173
- [Background] Chor J, Bregand-White J, Golobof A, Harwood B, Cowett A. Ibuprofen prophylaxis for levonorgestrel-releasing intrauterine system insertion: a randomized controlled trial. Contraception. 2012 Jun;85(6):558-62. doi: 10.1016/j.contraception.2011.10.015. Epub 2011 Dec 15. PMID 22176793
- [Background] Winner B, Peipert JF, Zhao Q, Buckel C, Madden T, Allsworth JE, Secura GM. Effectiveness of long-acting reversible contraception. N Engl J Med. 2012 May 24;366(21):1998-2007. doi: 10.1056/NEJMoa1110855. PMID 22621627
- [Background] Edelman AB, Schaefer E, Olson A, Van Houten L, Bednarek P, Leclair C, Jensen JT. Effects of prophylactic misoprostol administration prior to intrauterine device insertion in nulliparous women. Contraception. 2011 Sep;84(3):234-9. doi: 10.1016/j.contraception.2011.01.016. Epub 2011 Mar 3. PMID 21843686
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Background] Dijkhuizen K, Dekkers OM, Holleboom CA, de Groot CJ, Hellebrekers BW, van Roosmalen GJ, Janssen CA, Helmerhorst FM. Vaginal misoprostol prior to insertion of an intrauterine device: an RCT. Hum Reprod. 2011 Feb;26(2):323-9. doi: 10.1093/humrep/deq348. Epub 2010 Dec 15. PMID 21159683
- [Background] Heikinheimo O, Inki P, Kunz M, Parmhed S, Anttila AM, Olsson SE, Hurskainen R, Gemzell-Danielsson K. Double-blind, randomized, placebo-controlled study on the effect of misoprostol on ease of consecutive insertion of the levonorgestrel-releasing intrauterine system. Contraception. 2010 Jun;81(6):481-6. doi: 10.1016/j.contraception.2010.01.020. Epub 2010 Mar 1. PMID 20472114
- [Background] Talamo G, Liao J, Bayerl MG, Claxton DF, Zangari M. Oral administration of analgesia and anxiolysis for pain associated with bone marrow biopsy. Support Care Cancer. 2010 Mar;18(3):301-5. doi: 10.1007/s00520-009-0652-0. Epub 2009 May 21. PMID 19455356
- [Background] Park SH, Bang SM, Nam E, Cho EK, Shin DB, Lee JH, Ahn JY. A randomized double-blind placebo-controlled study of low-dose intravenous Lorazepam to reduce procedural pain during bone marrow aspiration and biopsy. Pain Med. 2008 Mar;9(2):249-52. doi: 10.1111/j.1526-4637.2006.00284.x. PMID 18298709
- [Background] Saav I, Aronsson A, Marions L, Stephansson O, Gemzell-Danielsson K. Cervical priming with sublingual misoprostol prior to insertion of an intrauterine device in nulliparous women: a randomized controlled trial. Hum Reprod. 2007 Oct;22(10):2647-52. doi: 10.1093/humrep/dem244. Epub 2007 Jul 25. PMID 17652452
- [Background] Davey HM, Barratt AL, Butow PN, Deeks JJ. A one-item question with a Likert or Visual Analog Scale adequately measured current anxiety. J Clin Epidemiol. 2007 Apr;60(4):356-60. doi: 10.1016/j.jclinepi.2006.07.015. Epub 2006 Dec 27. PMID 17346609
- [Background] Preutthipan S, Herabutya Y. A randomized comparison of vaginal misoprostol and dinoprostone for cervical priming in nulliparous women before operative hysteroscopy. Fertil Steril. 2006 Oct;86(4):990-4. doi: 10.1016/j.fertnstert.2006.03.039. Epub 2006 Sep 1. PMID 16949590
- [Background] Murty J. Use and effectiveness of oral analgesia when fitting an intrauterine device. J Fam Plann Reprod Health Care. 2003 Jul;29(3):150-1. doi: 10.1783/147118903101197539. PMID 12885310
- [Background] Wiebe E, Podhradsky L, Dijak V. The effect of lorazepam on pain and anxiety in abortion. Contraception. 2003 Mar;67(3):219-21. doi: 10.1016/s0010-7824(02)00516-4. PMID 12618257
- [Background] Kuganeswaran E, Clarkston WK, Cuddy PG, Quiason SG, Pandya PK, Dierenfeldt WT, Jonnalagadda SS, Smith OJ, Chen ST. A double-blind placebo controlled trial of oral midazolam as premedication before flexible sigmoidoscopy. Am J Gastroenterol. 1999 Nov;94(11):3215-9. doi: 10.1111/j.1572-0241.1999.01521.x. PMID 10566717
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419